CLINICAL TRIAL: NCT01240902
Title: Medtronic CoreValve® U.S. Pivotal Trial
Brief Title: Safety and Efficacy Study of the Medtronic CoreValve® System in the Treatment of Symptomatic Severe Aortic Stenosis in High Risk and Very High Risk Subjects Who Need Aortic Valve Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCV-US-2009-01
Record Dates: First submitted 2010-11-10; First posted 2010-11-15 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Severe Aortic Stenosis
Keywords: Valvular Heart Disease; Critical Aortic Stenosis; Severe Aortic Stenosis; High Risk; Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Extreme Risk: TAVI Iliofemoral (Experimental): Extreme Risk Patients: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI); Iliofemoral Access
  Interventions: Device: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
- Extreme Risk: TAVI Non-Iliofemoral (Experimental): Extreme Risk Patients: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI); Non-Iliofemoral Access
  Interventions: Device: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
- High Risk: TAVI (Experimental): High Risk Surgical Patients: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
  Interventions: Device: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
- High Risk: SAVR (Active Comparator): High Risk Surgical Patients: Surgical Aortic Valve Replacement (SAVR)
  Interventions: Device: Surgical Aortic Valve Replacement (SAVR)

INTERVENTIONS:
Device: Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI) — Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI)
  Arms: Extreme Risk: TAVI Iliofemoral; Extreme Risk: TAVI Non-Iliofemoral; High Risk: TAVI
Device: Surgical Aortic Valve Replacement (SAVR) — Surgical Aortic Valve Replacement (SAVR)
  Arms: High Risk: SAVR

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of the Medtronic CoreValve® System in the treatment of symptomatic severe aortic stenosis in subjects who have a predicted high risk for aortic valve surgery and/or very high risk for aortic valve surgery.

ELIGIBILITY:
Inclusion Criteria:

* Extreme Risk Only: Subject must have comorbidities such that one cardiologist and two cardiac surgeons agree that medical factors preclude operation, based on a conclusion that the probability of death or serious morbidity exceeds the probability of meaningful improvement. Specifically, the predicted operative risk of death or serious, irreversible morbidity is ≥ 50% at 30 days.
* High Risk Surgical Only: Subject must have comorbidities such that one cardiologist and two cardiac surgeons agree that predicted risk of operative mortality is ≥15% (and predicted operative mortality or serious, irreversible morbidity risk of < 50%) at 30 days.
* Subject has senile degenerative aortic valve stenosis with: mean gradient > 40 mmHg, or jet velocity greater than 4.0 m/sec by either resting or dobutamine stress echocardiogram, or simultaneous pressure recordings at cardiac catheterization (either resting or dobutamine stress), AND an initial aortic valve area of ≤ 0.8 cm2 (or aortic valve area index ≤ 0.5 cm2/m2) by resting echocardiogram or simultaneous pressure recordings at cardiac catheterization
* Subject is symptomatic from his/her aortic valve stenosis, as demonstrated by New York Heart Association (NYHA) Functional Class II or greater.
* The subject or the subject's legal representative has been informed of the nature of the trial, agrees to its provisions and has provided written informed consent as approved by the IRB of the respective clinical site.
* The subject and the treating physician agree that the subject will return for all required post-procedure follow-up visits.

Exclusion Criteria:

Clinical

* Evidence of an acute myocardial infarction ≤ 30 days before the intended treatment.
* Any percutaneous coronary or peripheral interventional procedure performed within 30 days prior to the intended treatment. (High Risk Surgical Only: Including bare metal stents. Additionally, any drug eluting stents placed within 6 months prior to the index procedure.)
* Blood dyscrasias as defined: leukopenia (WBC < 1000mm3), thrombocytopenia (platelet count <50,000 cells/mm3), history of bleeding diathesis or coagulopathy.
* Untreated clinically significant coronary artery disease requiring revascularization.
* Cardiogenic shock manifested by low cardiac output, vasopressor dependence, or mechanical hemodynamic support.
* Need for emergency surgery for any reason.
* Severe ventricular dysfunction with left ventricular ejection fraction (LVEF) < 20% as measured by resting echocardiogram.
* Recent (within 6 months) cerebrovascular accident (CVA) or transient ischemic attack (TIA).
* End stage renal disease requiring chronic dialysis or creatinine clearance < 20 cc/min.
* Active Gastrointestinal (GI) bleeding within the past 3 months.
* A known hypersensitivity or contraindication to any of the following which cannot be adequately pre-medicated:
* Aspirin
* Heparin (HIT/HITTS)
* Bivalirudin (Extreme Risk Only)
* Nitinol (titanium or nickel)
* Ticlopidine and clopidogrel
* Contrast media
* Ongoing sepsis, including active endocarditis.
* Subject refuses a blood transfusion.
* Life expectancy < 12 months due to associated non-cardiac co-morbid conditions.
* Other medical, social, or psychological conditions that in the opinion of an Investigator precludes the subject from appropriate consent.
* Severe dementia (resulting in either inability to provide informed consent for the trial/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits).
* Currently participating in an investigational drug or another device trial.
* Symptomatic carotid or vertebral artery disease.
* Subject has been offered surgical aortic valve replacement but declined. (High Risk Surgical Only)

Anatomical

* Native aortic annulus size < 18 mm or > 29 mm per the baseline diagnostic imaging.
* Pre-existing prosthetic heart valve any position.
* Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation (3-4+)).
* Moderate to severe (3-4+) or severe (4+) mitral or severe (4+) tricuspid regurgitation.
* Moderate to severe mitral stenosis.
* Hypertrophic obstructive cardiomyopathy.
* New or untreated echocardiographic evidence of intracardiac mass, thrombus or vegetation.
* Severe basal septal hypertrophy with an outflow gradient.
* Aortic root angulation (angle between plane of aortic valve annulus and horizontal plane/vertebrae) > 70° (for femoral and left subclavian/axillary access) and > 30° (for right subclavian/axillary access).
* Ascending aorta diameter > 43 mm if the aortic annulus diameter is 23-29 mm; ascending aorta diameter > 40 mm if the aortic annulus diameter is 20-23 mm; or an ascending aorta diameter > 34 mm if the aortic annulus diameter is 18-20 mm.
* Congenital bicuspid or unicuspid valve verified by echocardiography.
* Sinus of valsalva anatomy that would prevent adequate coronary perfusion.

Vascular

- Transarterial access not able to accommodate an 18Fr sheath.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1453 (Actual)
Dates: Start 2010-12-10 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Adams, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (45):
- United States (45):
  - Banner Good Samaritan, Phoenix, Arizona
  - Kaiser Permanente - Los Angeles Medical Center, Los Angeles, California
  - University of Southern California University Hospital, Los Angeles, California
  - El Camino Hospital, Mountain View, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Washington Hospital Center / Georgetown Hospital, Washington D.C., District of Columbia
  - University of Miami Health System / Jackson Memorial Hospital, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - Iowa Heart Center, Des Moines, Iowa
  - University of Kansas Hospital, Kansas City, Kansas
  - Cardiovascular Institute of the South/ Terrebone General, Houma, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Detroit Medical Center Cardiovascular Institute, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Morristown Memorial Hospital, Morristown, New Jersey
  - North Shore University Hospital/ Long Island Jewish Hospital, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - The Mount Sinai Medical Center, New York, New York
  - Lenox Hill Hospital, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University - Baptist Medical Center, Winston-Salem, North Carolina
  - University Hospitals - Case Medical Center, Cleveland, Ohio
  - The Ohio State University Medical Center - The Richard M. Ross Heart Hospital, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Pinnacle Health, Harrisburg, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - Texas Heart Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - The Methodist Hospital - The Methodist DeBakey Heart & Vascular Center, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - St. Luke's Medical Center - Aurora Health Care, Milwaukee, Wisconsin

REFERENCES:
- [Derived] O'Hair D, Yakubov SJ, Grubb KJ, Oh JK, Ito S, Deeb GM, Van Mieghem NM, Adams DH, Bajwa T, Kleiman NS, Chetcuti S, Sondergaard L, Gada H, Mumtaz M, Heiser J, Merhi WM, Petrossian G, Robinson N, Tang GHL, Rovin JD, Little SH, Jain R, Verdoliva S, Hanson T, Li S, Popma JJ, Reardon MJ. Structural Valve Deterioration After Self-Expanding Transcatheter or Surgical Aortic Valve Implantation in Patients at Intermediate or High Risk. JAMA Cardiol. 2023 Feb 1;8(2):111-119. doi: 10.1001/jamacardio.2022.4627. PMID 36515976
- [Derived] Lanz J, Reardon MJ, Pilgrim T, Stortecky S, Deeb GM, Chetcuti S, Yakubov SJ, Gleason TG, Huang J, Windecker S. Incidence and Outcomes of Infective Endocarditis After Transcatheter or Surgical Aortic Valve Replacement. J Am Heart Assoc. 2021 Oct 5;10(19):e020368. doi: 10.1161/JAHA.120.020368. Epub 2021 Sep 28. PMID 34581194
- [Derived] Arnold SV, Petrossian G, Reardon MJ, Kleiman NS, Yakubov SJ, Wang K, Hermiller J Jr, Harrison JK, Deeb GM, Huang J, Cohen DJ; US CoreValve Investigators. Five-Year Clinical and Quality of Life Outcomes From the CoreValve US Pivotal Extreme Risk Trial. Circ Cardiovasc Interv. 2021 Jun;14(6):e010258. doi: 10.1161/CIRCINTERVENTIONS.120.010258. Epub 2021 Jun 7. PMID 34092091
- [Derived] Arnold SV, Chinnakondepalli KM, Magnuson EA, Reardon MJ, Deeb GM, Gleason T, Yakubov SJ, Cohen DJ; CoreValve US Pivotal Trial Investigators. Five-Year Health Status After Self-expanding Transcatheter or Surgical Aortic Valve Replacement in High-risk Patients With Severe Aortic Stenosis. JAMA Cardiol. 2021 Jan 1;6(1):97-101. doi: 10.1001/jamacardio.2020.4397. PMID 32997095
- [Derived] Ito S, Nkomo VT, Orsinelli DA, Lin G, Cavalcante J, Popma JJ, Adams DH, Checuti SJ, Deeb GM, Boulware M, Huang J, Little SH, Cohen SA, Reardon MJ, Oh JK. Impact of Stroke Volume Index and Left Ventricular Ejection Fraction on Mortality After Aortic Valve Replacement. Mayo Clin Proc. 2020 Jan;95(1):69-76. doi: 10.1016/j.mayocp.2019.10.031. PMID 31902431
- [Derived] Lindman BR, Goel K, Bermejo J, Beckman J, O'Leary J, Barker CM, Kaiser C, Cavalcante JL, Elmariah S, Huang J, Hickey GL, Adams DH, Popma JJ, Reardon MJ. Lower Blood Pressure After Transcatheter or Surgical Aortic Valve Replacement is Associated with Increased Mortality. J Am Heart Assoc. 2019 Nov 5;8(21):e014020. doi: 10.1161/JAHA.119.014020. Epub 2019 Oct 31. PMID 31665959
- [Derived] Pineda AM, Kevin Harrison J, Kleiman NS, Reardon MJ, Conte JV, O'Hair DP, Chetcuti SJ, Huang J, Yakubov SJ, Popma JJ, Beohar N. Clinical impact of baseline chronic kidney disease in patients undergoing transcatheter or surgical aortic valve replacement. Catheter Cardiovasc Interv. 2019 Mar 1;93(4):740-748. doi: 10.1002/ccd.27928. Epub 2018 Oct 20. PMID 30341970
- [Derived] Gleason TG, Reardon MJ, Popma JJ, Deeb GM, Yakubov SJ, Lee JS, Kleiman NS, Chetcuti S, Hermiller JB Jr, Heiser J, Merhi W, Zorn GL 3rd, Tadros P, Robinson N, Petrossian G, Hughes GC, Harrison JK, Conte JV, Mumtaz M, Oh JK, Huang J, Adams DH; CoreValve U.S. Pivotal High Risk Trial Clinical Investigators. 5-Year Outcomes of Self-Expanding Transcatheter Versus Surgical Aortic Valve Replacement in High-Risk Patients. J Am Coll Cardiol. 2018 Dec 4;72(22):2687-2696. doi: 10.1016/j.jacc.2018.08.2146. Epub 2018 Sep 21. PMID 30249462
- [Derived] Grayburn PA, Oh JK, Reardon MJ, Popma JJ, Deeb GM, Boulware M, Huang J, Stoler RC. Effect of Baseline Aortic Regurgitation on Mortality in Patients Treated With Transcatheter or Surgical Aortic Valve Replacement (from the CoreValve US Pivotal Trial). Am J Cardiol. 2018 Nov 1;122(9):1527-1535. doi: 10.1016/j.amjcard.2018.07.018. Epub 2018 Aug 3. PMID 30172363
- [Derived] Crestanello JA, Popma JJ, Adams DH, Deeb GM, Mumtaz M, George B, Huang J, Reardon MJ. Long-Term Health Benefit of Transcatheter Aortic Valve Replacement in Patients With Chronic Lung Disease. JACC Cardiovasc Interv. 2017 Nov 27;10(22):2283-2293. doi: 10.1016/j.jcin.2017.07.025. Epub 2017 Nov 1. PMID 29102579
- [Derived] Kleiman NS, Maini BJ, Reardon MJ, Conte J, Katz S, Rajagopal V, Kauten J, Hartman A, McKay R, Hagberg R, Huang J, Popma J; CoreValve Investigators. Neurological Events Following Transcatheter Aortic Valve Replacement and Their Predictors: A Report From the CoreValve Trials. Circ Cardiovasc Interv. 2016 Sep;9(9):e003551. doi: 10.1161/CIRCINTERVENTIONS.115.003551. PMID 27601429
- [Derived] Reardon MJ, Kleiman NS, Adams DH, Yakubov SJ, Coselli JS, Deeb GM, O'Hair D, Gleason TG, Lee JS, Hermiller JB Jr, Chetcuti S, Heiser J, Merhi W, Zorn GL 3rd, Tadros P, Robinson N, Petrossian G, Hughes GC, Harrison JK, Maini B, Mumtaz M, Conte JV, Resar JR, Aharonian V, Pfeffer T, Oh JK, Huang J, Popma JJ. Outcomes in the Randomized CoreValve US Pivotal High Risk Trial in Patients With a Society of Thoracic Surgeons Risk Score of 7% or Less. JAMA Cardiol. 2016 Nov 1;1(8):945-949. doi: 10.1001/jamacardio.2016.2257. PMID 27541162
- [Derived] Popma JJ, Reardon MJ, Yakubov SJ, Hermiller JB Jr, Harrison JK, Gleason TG, Conte JV, Deeb GM, Chetcuti S, Oh JK, Boulware MJ, Huang J, Adams DH; CoreValve US Clinical Investigators. Safety and Efficacy of Self-Expanding TAVR in Patients With Aortoventricular Angulation. JACC Cardiovasc Imaging. 2016 Aug;9(8):973-81. doi: 10.1016/j.jcmg.2016.06.002. PMID 27491485
- [Derived] Hermiller JB Jr, Yakubov SJ, Reardon MJ, Deeb GM, Adams DH, Afilalo J, Huang J, Popma JJ; CoreValve United States Clinical Investigators. Predicting Early and Late Mortality After Transcatheter Aortic Valve Replacement. J Am Coll Cardiol. 2016 Jul 26;68(4):343-52. doi: 10.1016/j.jacc.2016.04.057. PMID 27443429
- [Derived] Popma JJ, Gleason TG, Yakubov SJ, Harrison JK, Forrest JK, Maini B, Ruiz CE, Pinto DS, Costa M, Resar J, Conte J, Crestanello J, Chang Y, Oh JK, Reardon MJ, Adams DH. Relationship of Annular Sizing Using Multidetector Computed Tomographic Imaging and Clinical Outcomes After Self-Expanding CoreValve Transcatheter Aortic Valve Replacement. Circ Cardiovasc Interv. 2016 Jul;9(7):e003282. doi: 10.1161/CIRCINTERVENTIONS.115.003282. PMID 27369803
- [Derived] Little SH, Oh JK, Gillam L, Sengupta PP, Orsinelli DA, Cavalcante JL, Chang JD, Adams DH, Zorn GL 3rd, Pollak AW, Abdelmoneim SS, Reardon MJ, Qiao H, Popma JJ. Self-Expanding Transcatheter Aortic Valve Replacement Versus Surgical Valve Replacement in Patients at High Risk for Surgery: A Study of Echocardiographic Change and Risk Prediction. Circ Cardiovasc Interv. 2016 Jun;9(6):e003426. doi: 10.1161/CIRCINTERVENTIONS.115.003426. PMID 27313280
- [Derived] Dauerman HL, Reardon MJ, Popma JJ, Little SH, Cavalcante JL, Adams DH, Kleiman NS, Oh JK. Early Recovery of Left Ventricular Systolic Function After CoreValve Transcatheter Aortic Valve Replacement. Circ Cardiovasc Interv. 2016 Jun;9(6):e003425. doi: 10.1161/CIRCINTERVENTIONS.115.003425. PMID 27296201
- [Derived] Deeb GM, Reardon MJ, Chetcuti S, Patel HJ, Grossman PM, Yakubov SJ, Kleiman NS, Coselli JS, Gleason TG, Lee JS, Hermiller JB Jr, Heiser J, Merhi W, Zorn GL 3rd, Tadros P, Robinson N, Petrossian G, Hughes GC, Harrison JK, Maini B, Mumtaz M, Conte J, Resar J, Aharonian V, Pfeffer T, Oh JK, Qiao H, Adams DH, Popma JJ; CoreValve US Clinical Investigators. 3-Year Outcomes in High-Risk Patients Who Underwent Surgical or Transcatheter Aortic Valve Replacement. J Am Coll Cardiol. 2016 Jun 7;67(22):2565-74. doi: 10.1016/j.jacc.2016.03.506. Epub 2016 Apr 3. PMID 27050187
- [Derived] Reynolds MR, Lei Y, Wang K, Chinnakondepalli K, Vilain KA, Magnuson EA, Galper BZ, Meduri CU, Arnold SV, Baron SJ, Reardon MJ, Adams DH, Popma JJ, Cohen DJ; CoreValve US High Risk Pivotal Trial Investigators. Cost-Effectiveness of Transcatheter Aortic Valve Replacement With a Self-Expanding Prosthesis Versus Surgical Aortic Valve Replacement. J Am Coll Cardiol. 2016 Jan 5;67(1):29-38. doi: 10.1016/j.jacc.2015.10.046. PMID 26764063
- [Derived] Oh JK, Little SH, Abdelmoneim SS, Reardon MJ, Kleiman NS, Lin G, Bach D, Gillam L, Kar B, Coselli J, Sengupta PP, Grewal K, Chang J, Chang Y, Boulware M, Adams DH, Popma JJ; CoreValve U.S. Pivotal Trial Clinical Investigators. Regression of Paravalvular Aortic Regurgitation and Remodeling of Self-Expanding Transcatheter Aortic Valve: An Observation From the CoreValve U.S. Pivotal Trial. JACC Cardiovasc Imaging. 2015 Dec;8(12):1364-1375. doi: 10.1016/j.jcmg.2015.07.012. Epub 2015 Oct 26. PMID 26508386
- [Derived] Yakubov SJ, Adams DH, Watson DR, Reardon MJ, Kleiman NS, Heimansohn D, Hermiller J Jr, Hughes GC, Harrison JK, Coselli J, Diez J, Schreiber T, Gleason TG, Conte J, Deeb GM, Huang J, Oh J, Byrne T, Caskey M, Popma JJ; CoreValve United States Clinical Investigators. 2-Year Outcomes After Iliofemoral Self-Expanding Transcatheter Aortic Valve Replacement in Patients With Severe Aortic Stenosis Deemed Extreme Risk for Surgery. J Am Coll Cardiol. 2015 Sep 22;66(12):1327-34. doi: 10.1016/j.jacc.2015.07.042. PMID 26383718
- [Derived] Arnold SV, Reynolds MR, Wang K, Magnuson EA, Baron SJ, Chinnakondepalli KM, Reardon MJ, Tadros PN, Zorn GL, Maini B, Mumtaz MA, Brown JM, Kipperman RM, Adams DH, Popma JJ, Cohen DJ; CoreValve US Pivotal Trial Investigators. Health Status After Transcatheter or Surgical Aortic Valve Replacement in Patients With Severe Aortic Stenosis at Increased Surgical Risk: Results From the CoreValve US Pivotal Trial. JACC Cardiovasc Interv. 2015 Aug 17;8(9):1207-1217. doi: 10.1016/j.jcin.2015.04.018. PMID 26292584
- [Derived] Reardon MJ, Adams DH, Kleiman NS, Yakubov SJ, Coselli JS, Deeb GM, Gleason TG, Lee JS, Hermiller JB Jr, Chetcuti S, Heiser J, Merhi W, Zorn GL 3rd, Tadros P, Robinson N, Petrossian G, Hughes GC, Harrison JK, Maini B, Mumtaz M, Conte JV, Resar JR, Aharonian V, Pfeffer T, Oh JK, Qiao H, Popma JJ. 2-Year Outcomes in Patients Undergoing Surgical or Self-Expanding Transcatheter Aortic Valve Replacement. J Am Coll Cardiol. 2015 Jul 14;66(2):113-21. doi: 10.1016/j.jacc.2015.05.017. Epub 2015 Jun 5. PMID 26055947
- [Derived] Osnabrugge RL, Arnold SV, Reynolds MR, Magnuson EA, Wang K, Gaudiani VA, Stoler RC, Burdon TA, Kleiman N, Reardon MJ, Adams DH, Popma JJ, Cohen DJ; CoreValve U.S. Trial Investigators. Health status after transcatheter aortic valve replacement in patients at extreme surgical risk: results from the CoreValve U.S. trial. JACC Cardiovasc Interv. 2015 Feb;8(2):315-323. doi: 10.1016/j.jcin.2014.08.016. PMID 25700755
- [Derived] Reardon MJ, Adams DH, Coselli JS, Deeb GM, Kleiman NS, Chetcuti S, Yakubov SJ, Heimansohn D, Hermiller J Jr, Hughes GC, Harrison JK, Khabbaz K, Tadros P, Zorn GL 3rd, Merhi W, Heiser J, Petrossian G, Robinson N, Maini B, Mumtaz M, Lee JS, Gleason TG, Resar J, Conte J, Watson D, Chenoweth S, Popma JJ; CoreValve US Clinical Investigators. Self-expanding transcatheter aortic valve replacement using alternative access sites in symptomatic patients with severe aortic stenosis deemed extreme risk of surgery. J Thorac Cardiovasc Surg. 2014 Dec;148(6):2869-76.e1-7. doi: 10.1016/j.jtcvs.2014.07.020. Epub 2014 Jul 30. PMID 25152474
- [Derived] Adams DH, Popma JJ, Reardon MJ, Yakubov SJ, Coselli JS, Deeb GM, Gleason TG, Buchbinder M, Hermiller J Jr, Kleiman NS, Chetcuti S, Heiser J, Merhi W, Zorn G, Tadros P, Robinson N, Petrossian G, Hughes GC, Harrison JK, Conte J, Maini B, Mumtaz M, Chenoweth S, Oh JK; U.S. CoreValve Clinical Investigators. Transcatheter aortic-valve replacement with a self-expanding prosthesis. N Engl J Med. 2014 May 8;370(19):1790-8. doi: 10.1056/NEJMoa1400590. Epub 2014 Mar 29. PMID 24678937
- [Derived] Popma JJ, Adams DH, Reardon MJ, Yakubov SJ, Kleiman NS, Heimansohn D, Hermiller J Jr, Hughes GC, Harrison JK, Coselli J, Diez J, Kafi A, Schreiber T, Gleason TG, Conte J, Buchbinder M, Deeb GM, Carabello B, Serruys PW, Chenoweth S, Oh JK; CoreValve United States Clinical Investigators. Transcatheter aortic valve replacement using a self-expanding bioprosthesis in patients with severe aortic stenosis at extreme risk for surgery. J Am Coll Cardiol. 2014 May 20;63(19):1972-81. doi: 10.1016/j.jacc.2014.02.556. Epub 2014 Mar 19. PMID 24657695

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between Feb 17, 2011 and Aug 23, 2013, 656 subjects were enrolled into the CoreValve US Pivotal Trial Extreme Risk study at 41 of the 43 activated centers in the United States. Between February 2, 2011 and July 23, 2013, 797 subjects were enrolled into the CoreValve US Pivotal Trial High Risk study at 45 centers in the United States.
Pre-assignment Details: The first 3 successfully enrolled and implanted iliofemoral subjects at each implanting site, inclusive of both the High Risk Surgical and Extreme Risk patient populations were considered roll-in subjects, and were automatically assigned to undergo Medtronic CoreValve® System Transcatheter Aortic Valve Implantation (TAVI).
Period: Overall Study
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Started | 500 | 156 | 395 | 402
Completed | 289 | 77 | 295 | 237
Not Completed | 211 | 79 | 100 | 165

BASELINE CHARACTERISTICS:
Population: Participant Population= As Treated (AT) cohort. The AT cohort consisted of all Intent to Treat (ITT) subjects with an attempted implant procedure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR | Total
Number analyzed (Participants) | 489 | 150 | 391 | 359 | 1389
Age, Continuous [Mean (Standard Deviation); unit: years] — Participant Population= Consisted of all subjects with an attempted implant procedure.
  years | 83.2 (8.7) | 81.3 (7.4) | 83.2 (7.1) | 83.3 (6.4) | 83.0 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Participant Population= Consisted of all subjects with an attempted implant procedure.
  Participants
    Female | 255 | 82 | 184 | 171 | 692
    Male | 234 | 68 | 207 | 188 | 697
Race/Ethnicity, Customized [Number; unit: participants] — Participant Population= Consisted of all subjects with an attempted implant procedure.
  participants
    American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
    Asian | 2 | 1 | 0 | 1 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 19 | 5 | 3 | 11 | 38
    White | 468 | 143 | 387 | 343 | 1341
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 1 | 1 | 2 | 4
Body Surface Area [Mean (Standard Deviation); unit: m^2] — Participant Population= Consisted of all subjects with an attempted implant procedure.
  m^2 | 1.8 (0.3) | 1.8 (0.2) | 1.8 (0.2) | 1.9 (0.2) | 1.8 (0.2)
NYHA Classification [Number; unit: participants] — New York Heart Association (NYHA) Classification:
  Class I: Subjects with cardiac disease but without resulting limitations of physical activity.
  Class I: Subjects with cardiac disease resulting in slight limitation of physical activity.
  Class III: Subjects with cardiac disease resulting in marked limitation of physical activity.
  Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort.
  participants
    NYHA I | 0 | 0 | 0 | 0 | 0
    NYHA II | 40 | 12 | 57 | 47 | 156
    NYHA III | 313 | 98 | 255 | 250 | 916
    NYHA IV | 136 | 40 | 79 | 62 | 317
Society of Thoracic Surgeons (STS) Risk Score [Mean (Standard Deviation); unit: % risk of mortality or morbidity] — The Society of Thoracic Surgeons (STS) risk model predicts the risk of operative mortality and morbidity after adult cardiac surgery on the basis of patient demographic and clinical variables. After information has been entered on a given case, the online STS risk calculator provides a risk percentage for each of the outcomes. The risk percentage estimates the chance of a specific outcome for a patient with the indicated risk factors. A higher score indicates a higher risk. A lower score indicates a lower risk.
  % risk of mortality or morbidity | 10.3 (5.5) | 10.7 (5.7) | 7.3 (3.0) | 7.5 (3.3) | 8.8 (4.7)
Logistic European System for Cardiac Operative Risk Evaluation (EuroSCORE) [Mean (Standard Deviation); unit: %] — The European System for Cardiac Operative Risk Evaluation (EuroSCORE) is a method of calculating predicted operative mortality for patients undergoing cardiac surgery. If a risk factor is present, a weight/number is assigned. The weights are added to give an approximate percent of predicted mortality. A higher score indicates a higher risk. A lower score indicates a lower risk.
  % | 22.6 (17.1) | 22.9 (15.9) | 17.7 (13.0) | 18.8 (13.2) | 20.3 (15.1)

OUTCOME MEASURES:

1. Primary Outcome: Extreme Risk: All-cause Death or Major Stroke; High Risk Surgical: All-cause Mortality
Description: All-cause Death or Major Stroke (Extreme Risk- Medtronic CoreValve® System); All-cause Mortality (High Risk Surgical- Medtronic CoreValve® System vs. Surgical Valve)
Time Frame: 1 year
Population: Participant Population= Consisted of all subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants, Kaplan-Meier
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 489 | 150 | 391 | 359
percentage of participants, Kaplan-Meier | 26.0 | 39.3 | 14.1 | 18.9
Statistical Analysis 1: Comparison: Extreme Risk: TAVI Iliofemoral; TAVR with the Medtronic CoreValve System meets the Performance Goal in the 12 month rate of all-cause mortality or major stroke H0: = πMCS TAVI ≥ 43.0% HA: = πMCS TAVI < 43.0% In the above expressions πMCS TAVI denotes the rate of all-cause mortality or major stroke during a fixed follow-up of 1 year; Test type: Superiority or Other; p < 0.0001, z-test, 1 sided; Kaplan-Meier = 26.0, 95% CI 2-sided [22.3 to 30.1], Standard Error of Mean 2.0 — Kaplan-Meier Event Rate Greenwood Standard Error
Statistical Analysis 2: Comparison: Extreme Risk: TAVI Non-Iliofemoral; No performance goal created, only descriptive statistics are provided; Test type: Superiority or Other; Kaplan-Meier = 39.3, Standard Error of Mean 4.0 — Kaplan-Meier Event Rate Greenwood Standard Error
Statistical Analysis 3: Comparison: High Risk: TAVI; Test type: Non-Inferiority or Equivalence — The 12 month all-cause mortality estimated rate was 20% for each group with a noninferiority margin of 7.5 percentage points. Assuming a 1:1 ratio in the treatment assignments, we estimated that a total of 355 patients were required in each group for the study to have power of 80% at a one-sided alpha level of 0.05. Accounting for a 10% loss to follow-up, we calculated that we would need to enroll 790 patients; p < 0.0001, z-test, 1 sided

2. Secondary Outcome: Major Adverse Cardiovascular and Cerebrovascular Event (MACCE)
Description: MACCE is defined as a composite of:
  * All Cause Mortality
  * Myocardial infarction (MI)
  * All Stroke
  * Reintervention (defined as any cardiac surgery or percutaneous reintervention catheter procedure that repairs, otherwise alters or adjusts, or replaces a previously implanted valve)
Time Frame: 30 day, 6 month, 1 year, 2 year
Population: Participant Population= Consisted of all subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants, Kaplan-Meier
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 489 | 150 | 391 | 359
percentage of participants, Kaplan-Meier
  30 day | 12.3 | 17.3 | 7.7 | 10.3
  6 month | 22.5 | 34.7 | 15.4 | 21.0
  1 year | 29.2 | 41.4 | 20.5 | 27.0
  2 Year | 42.3 | 51.0 | 29.7 | 38.6
Statistical Analysis 1: Comparison: High Risk: TAVI vs High Risk: SAVR; Powered Secondary Hypothesis: TAVR with the Medtronic CoreValve System was superior to SAVR in binary rate of MACCE at 30 days or hospital discharge, whichever was longer: H0: πMCS TAVR = πSAVR HA: πMCS TAVR < πSAVR In the above expression πMCS TAVR and πSAVR denoted rates of MACCE at 30 days or hospital discharge, whichever was longer. Assumptions: 1:1 treatment allocation ratio One-sided alpha=0.025 SAVR = 20.0% MCS TAVI = 12.1% Power = >80%; Test type: Superiority or Other; p = 0.1033, Kaplan-Meier Point Estimate — Hierarchical test item #5, MACCE at 30 days or hospital discharge; whichever was longer. K-M rates TAVR 8.21%, SAVR 10.93%, Difference -2.73%, Standard Error 2.16%, and Upper 95% CI 1.5%; Using Greenwood formula

3. Secondary Outcome: The Occurrence of Individual MACCE Components
Description: Individual MACCE Components Include:
  * All Cause Mortality
  * MI
  * All stroke
  * Reintervention (defined as any cardiac surgery or percutaneous reintervention catheter procedure that repairs, otherwise alters or adjusts, or replaces a previously implanted valve)
Time Frame: 30 day, 6 month, 1 year, 2 year
Population: Participant Population= Consisted of all subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants, Kaplan-Meier
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 489 | 150 | 391 | 359
percentage of participants, Kaplan-Meier
  30 day All Cause Mortality | 8.4 | 11.3 | 3.3 | 4.5
  30 day MI | 1.2 | 2.1 | 0.8 | 0.8
  30 day Stroke | 4.0 | 8.8 | 4.9 | 6.2
  30 day Reintervention | 1.1 | 0.0 | 0.8 | 0.0
  6 month All Cause Mortality | 18.6 | 28.7 | 9.0 | 14.0
  6 month MI | 1.5 | 2.1 | 1.6 | 1.1
  6 month Stroke | 5.2 | 12.0 | 7.3 | 9.9
  6 month Reintervention | 1.5 | 0.0 | 1.0 | 0.0
  1 year All Cause Mortality | 24.3 | 36.0 | 14.1 | 18.9
  1 year MI | 2.0 | 2.1 | 1.9 | 1.5
  1 year Stroke | 7.0 | 13.0 | 8.7 | 12.5
  1 year Reintervention | 1.8 | 1.0 | 2.2 | 0.0
  2 year All Cause Mortality | 36.6 | 44.9 | 22.2 | 28.6
  2 year MI | 2.8 | 3.2 | 1.9 | 2.3
  2 year Stroke | 8.6 | 16.1 | 10.9 | 16.6
  2 year Reintervention | 1.8 | 1.0 | 2.5 | 0.4

4. Secondary Outcome: Major Adverse Events (MAEs)
Description: MAEs Include:
  * MACCE
  * Acute Kidney Injury
  * Cardiac Tamponade
  * Prosthetic Valve Dysfunction
  * Cardiogenic Shock
  * Valve Endocarditis
  * Life-Threatening, Disabling or Major Bleeding
  * Major Vascular Complication
  * Cardiac Perforation
  * Device Migration/Valve Embolism
Time Frame: 30 day, 6 month, 1 year, 2 year
Population: Participant Population= Consisted of all subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants, Kaplan-Meier
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 489 | 150 | 391 | 359
percentage of participants, Kaplan-Meier
  30 day | 54.2 | 69.3 | 52.4 | 50.2
  6 month | 60.5 | 76.0 | 58.6 | 76.4
  1 year | 63.4 | 80.0 | 60.1 | 59.8
  2 year | 71.3 | 84.0 | 66.4 | 66.8

5. Secondary Outcome: Conduction Disturbance Requiring Permanent Pacemaker Implantation
Time Frame: 30 day, 6 month, 1 year, 2 year
Population: Participant Population= Consisted of all subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants, Kaplan-Meier
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 489 | 150 | 391 | 359
percentage of participants, Kaplan-Meier
  30 day | 21.6 | 16.4 | 20.0 | 7.1
  6 month | 24.4 | 20.5 | 21.9 | 9.9
  1 year | 26.4 | 21.5 | 22.5 | 11.6
  2 year | 28.8 | 22.6 | 25.8 | 12.8

6. Secondary Outcome: Change in NYHA Class
Description: Change from baseline (continuous variable). A positive number corresponds to NYHA worsening; a negative number corresponds to NYHA improvement.
  New York Heart Association (NYHA) Classification:
  Class I: Subjects with cardiac disease but without resulting limitations of physical activity.
  Class I: Subjects with cardiac disease resulting in slight limitation of physical activity.
  Class III: Subjects with cardiac disease resulting in marked limitation of physical activity.
  Class IV: Subjects with cardiac disease resulting in inability to carry on any physical activity without discomfort.
Time Frame: 30 day, 6 month, 1 year, 2 year
Population: Participant Population= Consisted of all subjects with an attempted implant procedure.
Measure: Mean (Standard Deviation); unit: average classification level change
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 489 | 150 | 391 | 359
average classification level change
  30 day | -1.3 (0.9) | -1.0 (0.8) | -1.3 (0.8) | -1.0 (0.9)
  6 month | -1.6 (0.9) | -1.4 (0.8) | -1.5 (0.8) | -1.4 (0.8)
  1 year | -1.6 (0.9) | -1.4 (0.8) | -1.5 (0.8) | -1.5 (0.8)
  2 year | -1.6 (0.8) | -1.4 (0.7) | -1.5 (0.8) | -1.5 (0.9)
Statistical Analysis 1: Comparison: Extreme Risk: TAVI Iliofemoral; Change in NYHA classification from baseline to 1 year from secondary objective #5. The paired t-test will be used to test the null hypothesis that the mean paired difference is zero versus the two-sided alternative that the mean is not zero; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Hierarchical test item #3, change from baseline to 1 year; Mean Difference (Net) = -1.6, Standard Deviation 0.9
Statistical Analysis 2: Comparison: High Risk: TAVI vs High Risk: SAVR; Change in NYHA classification from baseline to 1 year: TAVR vs. SAVR from secondary objective #5. The one-sided two-sample t-test was used to test non-inferiority at a level 0.05 the hypotheses: H0: µ MCS TAVR ≤ µ SAVR -0.375 HA: µ MCS TAVR > µ SAVR -0.375 In the above expression µ MCS TAVR and µ SAVR denoted the mean number of classification improvements in NYHA from baseline to 1 year; Test type: Non-Inferiority or Equivalence — Non-inferiority margin= 0.375. For subjects with NYHA categories at both baseline and 1 year visit, the NYHA classification improvements were calculated as NYHAbaseline - NYHA1year; p < 0.0001, t-test, 1 sided — Hierarchical test item #3, change from baseline to 1 year

7. Secondary Outcome: Change in Distance Walked During 6-Minute Walk Test (6MWT)
Description: Change in distance walked during 6MWT from baseline
Time Frame: 30 day, 1 year
Population: Participant Population= Consisted of all subjects with an attempted implant procedure.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 489 | 150 | 391 | 359
meters
  30 day | 19.6 (109.1) | 13.3 (110.0) | 25.8 (105.5) | -6.9 (89.8)
  1 year | 13.9 (140.4) | 22.2 (136.2) | 27.0 (114.3) | 24.0 (111.8)

8. Secondary Outcome: Ratio of Days Alive Out of Hospital Versus Total Days Alive
Time Frame: 1 year
Population: Participant Population= Consisted of all subjects with an attempted implant procedure.
Measure: Mean (Standard Deviation); unit: ratio of days alive and out of hospital
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 489 | 150 | 391 | 359
ratio of days alive and out of hospital | 0.86 (0.28) | 0.81 (0.31) | 0.92 (0.20) | 0.89 (0.23)

9. Secondary Outcome: Quality of Life (QoL) Change
Description: QoL summary score change from baseline using the following measures:
  * Kansas City Cardiomyopathy Questionnaire (KCCQ): Quantifies physical function, symptoms, social function, self-efficacy and knowledge, and quality of life. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
  * 12 Item Short Form Health Survey (SF-12): Measures functional health and well-being. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
  * European QoL (EQ-5D): Measures 5 domains (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) that can be converted to utilities using an algorithm. Utilities range from 0 to 1, with 1 representing perfect health, and 0 corresponding to the worst imaginable health state.
Time Frame: 30 day, 6 month, 1 year, 2 year
Population: Participant Population= Consisted of all subjects with an attempted implant procedure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 489 | 150 | 391 | 359
units on a scale
  30 day KCCQ- Overall | 24.2 (28.9) | 7.9 (33.5) | 19.0 (29.4) | 4.3 (28.1)
  30 day KCCQ- Clinical | 20.2 (28.0) | 6.8 (32.0) | 14.7 (28.6) | 2.7 (27.1)
  30 day SF-12-Physical | 5.9 (10.4) | 1.9 (10.4) | 4.9 (10.2) | -0.0 (10.1)
  30 day SF-12-Mental | 3.7 (14.2) | -1.7 (16.2) | 2.6 (13.1) | -2.5 (13.4)
  30 day EQ-5D | 0.09 (0.29) | 0.00 (0.30) | 0.04 (0.24) | -0.07 (0.26)
  6 month KCCQ-Overall | 27.4 (27.0) | 23.1 (28.3) | 24.8 (26.9) | 22.9 (26.4)
  6 month KCCQ- Clinical | 22.2 (26.1) | 17.5 (26.6) | 18.6 (25.7) | 17.7 (25.7)
  6 month SF-12-Physical | 5.2 (11.3) | 4.5 (8.9) | 6.3 (11.0) | 6.2 (9.9)
  6 month SF-12-Mental | 4.6 (13.6) | 4.4 (13.8) | 4.6 (11.8) | 2.6 (13.1)
  6 month EQ-5D | 0.09 (0.22) | 0.05 (0.21) | 0.05 (0.22) | 0.04 (0.17)
  1 year KCCQ-Overall | 27.9 (27.1) | 21.9 (26.8) | 23.2 (25.4) | 21.8 (26.5)
  1 year KCCQ- Clinical | 20.8 (26.8) | 18.1 (24.9) | 16.7 (25.5) | 15.2 (26.0)
  1 year SF-12-Physical | 5.5 (10.8) | 4.6 (10.0) | 6.0 (11.5) | 5.3 (10.3)
  1 year SF-12-Mental | 5.2 (13.7) | 2.4 (14.3) | 4.5 (11.8) | 3.2 (12.1)
  1 year EQ-5D | 0.06 (0.25) | 0.05 (0.25) | 0.04 (0.19) | 0.01 (0.19)
  2 year KCCQ - Overall | 25.2 (27.2) | 14.9 (29.5) | 22.2 (26.5) | 18.7 (25.6)
  2 year KCCQ - Clinical | 18.8 (26.1) | 11.6 (26.9) | 14.6 (26.0) | 12.6 (25.8)
  2 year SF-12 - Physical | 4.0 (11.2) | 1.9 (11.9) | 5.0 (12.1) | 4.3 (10.2)
  2 year SF-12 - Mental | 3.8 (15.3) | 2.2 (14.8) | 3.6 (13.0) | 1.7 (13.0)
  2 year EQ-5D | 0.04 (0.25) | 0.03 (0.26) | -0.01 (0.24) | -0.01 (0.21)
Statistical Analysis 1: Comparison: Extreme Risk: TAVI Iliofemoral; Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) score from baseline to 1 year from secondary objective #8. The paired t-test will be used to test the null hypothesis that the mean paired difference is zero versus the two-sided alternative that the mean is not zero; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Hierarchical test item #4
Statistical Analysis 2: Comparison: High Risk: TAVI vs High Risk: SAVR; Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) score from baseline to 1 year: TAVR vs. SAVR from secondary objective #8. The one-sided two-sample t-test was used to test non-inferiority at a level 0.05 the hypotheses: H0: µ MCS TAVR ≤ µ SAVR -5 HA: µ MCS TAVR > µ SAVR -5 In the above expression µ MCS TAVR and µ SAVR denoted the mean improvements in the KCCQ score from baseline to 1 year; Test type: Non-Inferiority or Equivalence — Non-inferiority margin 5; p = 0.0063, t-test, 1 sided — Hierarchical test item #4
Statistical Analysis 3: Comparison: High Risk: TAVI vs High Risk: SAVR; Change in SF-12 Physical Summary Scale from baseline to 30 days: TAVR vs. SAVR from secondary objective #8. The two-sided two-sample t-test was used to test at a level 0.05 the hypotheses: H0: µ MCS TAVR = µ SAVR HA: µ MCS TAVR ≠ µ SAVR In the above expression µ MCS TAVR and µ SAVR denoted the mean improvements in the SF-12 Physical Summary Scale from baseline to 30 days; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Hierarchical test item #6. Item #5 failed, therefore, item #6 also fails. Nominal p- value provided

10. Secondary Outcome: Echocardiographic Assessment of Valve Performance
Description: Using the following measures:
  - Effective Orifice Area (EOA)
Time Frame: 30 day, 6 month, 1 year, 2 year
Population: Participant Population= Consisted of all subjects with a valve implanted.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 486 | 148 | 390 | 354
cm^2
  30 day EOA | 1.86 (0.56) | 1.82 (0.64) | 1.94 (0.56) | 1.60 (0.51)
  6 month EOA | 1.88 (0.55) | 1.85 (0.51) | 1.91 (0.53) | 1.56 (0.49)
  1 year EOA | 1.88 (0.54) | 1.85 (0.51) | 1.91 (0.52) | 1.57 (0.49)
  2 year EOA | 1.86 (0.55) | 1.83 (0.58) | 1.87 (0.48) | 1.51 (0.43)
Statistical Analysis 1: Comparison: Extreme Risk: TAVI Iliofemoral; EOA: Change in effective orifice area from Baseline to 1 year from secondary objective #9. The paired t-test will be used to test the null hypothesis that the mean paired difference is zero versus the two-sided alternative that the mean is not zero; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Hierarchical test item #2
Statistical Analysis 2: Comparison: High Risk: TAVI vs High Risk: SAVR; EOA: Change in effective orifice area from Baseline to 1 year: TAVR vs.SAVR from secondary objective #9. The one-sided two-sample t-test was used to test non-inferiority at a level 0.05 the hypotheses: H0: µ MCS TAVR ≤ µ SAVR -0.375 HA: µ MCS TAVR > µ SAVR -0.375 In the above expression µ MCS TAVR and µ SAVR denoted the mean improvements in effective orifice area from Baseline to 1 year measured in cm2; Test type: Non-Inferiority or Equivalence — Non-inferiority margin 0.375; p < 0.0001, t-test, 1 sided — Hierarchical test item #2

11. Secondary Outcome: Echocardiographic Assessment of Valve Performance
Description: Using the following measures:
  - Transvalvular Mean Gradient
Time Frame: 30 day, 6 month, 1 year, 2 year
Population: Participant Population= Consisted of all subjects with a valve implanted.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 486 | 148 | 390 | 354
mmHg
  30 day Mean Gradient | 8.68 (4.16) | 9.74 (5.82) | 8.88 (3.86) | 11.72 (5.70)
  6 month Mean Gradient | 9.10 (3.89) | 9.42 (5.60) | 9.08 (4.08) | 12.12 (6.31)
  1 year Mean Gradient | 8.86 (4.09) | 9.46 (5.65) | 9.09 (3.49) | 12.44 (7.36)
  2 year Mean Gradient | 8.70 (4.22) | 9.24 (5.35) | 8.47 (3.76) | 12.05 (6.32)
Statistical Analysis 1: Comparison: Extreme Risk: TAVI Iliofemoral; Transvalvular Mean Gradient: Change in transvalvular mean gradient from baseline to 1 year from secondary objective #9. The paired t-test will be used to test the null hypothesis that the mean paired difference is zero versus the two-sided alternative that the mean is not zero; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Hierarchical test item #1
Statistical Analysis 2: Comparison: High Risk: TAVI vs High Risk: SAVR; Transvalvular Mean Gradient: Change in transvalvular mean gradient from baseline to 1 year: TAVR vs.SAVR from secondary objective #9. The one-sided two-sample t-test was used to test non-inferiority at a level of 0.05 the hypotheses: H0: μ MCS TAVR ≤ μ SAVR -15 HA: μ MCS TAVR > μ SAVR -15 In the above expression μ MCS TAVR and μ SAVR denoted the mean improvements in mean gradient from Baseline to 1 year measured in mmHg; Test type: Non-Inferiority or Equivalence — Non-inferiority margin 15; p < 0.0001, t-test, 1 sided — Hierarchical test item #1

12. Secondary Outcome: Echocardiographic Assessment of Valve Performance
Description: Using the following measure:
  - Degree of Aortic Valve Regurgitation (Transvalvular and Paravalvular)
Time Frame: 30 day, 6 month, 1 year, 2 year
Population: Participant Population= Consisted of all subjects with a valve implanted.
Measure: Number; unit: percentage of participants
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 486 | 148 | 390 | 354
percentage of participants
  30 day Total Aortic Regurgitation- None | 9.1 | 19.0 | 12.2 | 65.0
  30 day Total Aortic Regurgitation- Trivial | 32.7 | 33.9 | 41.4 | 23.0
  30 day Total Aortic Regurgitation- Mild | 43.0 | 34.7 | 36.4 | 10.7
  30 day Total Aortic Regurgitation- Moderate | 14.1 | 10.7 | 8.1 | 1.3
  30 day Total Aortic Regurgitation- Severe | 1.2 | 1.7 | 1.9 | 0.0
  6 month Total Aortic Regurgitation- None | 19.9 | 33.3 | 21.6 | 60.6
  6 month Total Aortic Regurgitation- Trivial | 33.5 | 27.1 | 37.2 | 28.0
  6 month Total Aortic Regurgitation- Mild | 36.5 | 35.4 | 29.7 | 9.8
  6 month Total Aortic Regurgitation- Moderate | 9.8 | 4.2 | 10.0 | 1.6
  6 month Total Aortic Regurgitation- Severe | 0.3 | 0.0 | 1.6 | 0.0
  1 year Total Aortic Regurgitation- None | 21.5 | 39.0 | 28.3 | 68.1
  1 year Total Aortic Regurgitation- Trivial | 40.6 | 36.6 | 35.7 | 21.7
  1 year Total Aortic Regurgitation- Mild | 31.5 | 20.7 | 29.0 | 8.8
  1 year Total Aortic Regurgitation- Moderate | 6.4 | 2.4 | 6.7 | 0.9
  1 year Total Aortic Regurgitation- Severe | 0.0 | 1.2 | 0.3 | 0.4
  2 year Total Aortic Regurgitation - None | 31.0 | 35.3 | 32.8 | 58.5
  2 year Total Aortic Regurgitation - Trivial | 26.3 | 36.8 | 27.0 | 27.3
  2 year Total Aortic Regurgitation - Mild | 36.1 | 23.5 | 32.0 | 13.1
  2 year Total Aortic Regurgitation - Moderate | 6.7 | 4.4 | 6.6 | 1.1
  2 year Total Aortic Regurgitation - Severe | 0.0 | 0.0 | 1.6 | 0.0

13. Secondary Outcome: Aortic Valve Hospitalizations
Time Frame: 30 day, 6 month, 1 year, 2 year
Population: Participant Population= Consisted of all subjects with an attempted implant procedure
Measure: Number; unit: percentage of participants, Kaplan-Meier
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 489 | 150 | 391 | 359
percentage of participants, Kaplan-Meier
  30 day | 6.7 | 8.7 | 3.9 | 5.2
  6 month | 16.4 | 18.3 | 13.4 | 9.0
  1 year | 21.9 | 21.2 | 16.5 | 14.0
  2 year | 29.5 | 27.2 | 24.2 | 18.2

14. Secondary Outcome: Cardiovascular Deaths and Valve Related Deaths
Time Frame: 30 day, 6 month, 1 year, 2 year
Population: Participant Population= Consisted of all subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants, Kaplan-Meier
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 489 | 150 | 391 | 359
percentage of participants, Kaplan-Meier
  30 day Cardiovascular Deaths | 8.4 | 11.3 | 3.3 | 4.5
  30 Day Valve Related Deaths | 2.5 | 2.8 | 2.3 | 0.6
  6 month Cardiovascular Deaths | 15.0 | 23.6 | 7.4 | 10.5
  6 month Valve Related Deaths | 4.1 | 4.5 | 3.6 | 1.8
  1 year Cardiovascular Deaths | 18.3 | 28.7 | 10.6 | 12.9
  1 year Valve Related Deaths | 5.1 | 5.4 | 5.6 | 2.2
  2 year Cardiovascular Deaths | 26.2 | 35.1 | 15.4 | 19.4
  2 year Valve Related Deaths | 6.2 | 7.5 | 6.8 | 4.2

15. Secondary Outcome: Strokes and Transient Ischemic Attacks (TIAs)
Description: Strokes (of any severity) and TIAs
Time Frame: 30 day, 6 month, 1 year, 2 year
Population: Participant Population= Consisted of all subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants, Kaplan-Meier
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 489 | 150 | 391 | 359
percentage of participants, Kaplan-Meier
  30 day | 4.6 | 10.2 | 5.7 | 6.5
  6 month | 6.0 | 14.3 | 8.4 | 10.8
  1 year | 8.1 | 15.2 | 10.3 | 14.1
  2 year | 10.1 | 19.5 | 13.2 | 17.8

16. Secondary Outcome: Index Procedure Related MAEs
Time Frame: Procedure
Population: Participant Population= Consisted of all subjects with an attempted implant procedure.
Measure: Number; unit: percentage of participants
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 489 | 150 | 391 | 359
percentage of participants | 53.5 | 68.9 | 52.6 | 49.9

17. Secondary Outcome: Length of Index Procedure Hospital Stay
Time Frame: Number of days from admission to discharge
Population: Participant Population= Consisted of all subjects with an attempted implant procedure.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 489 | 150 | 391 | 359
days | 9.2 (8.1) | 11.2 (8.9) | 8.0 (6.8) | 12.5 (10.7)

18. Secondary Outcome: Device Success
Description: Medtronic CoreValve® System subjects only.
  Defined as:
  * Successful vascular access, delivery and deployment of the device, and successful retrieval of the delivery system,
  * Correct position of the device in the proper anatomical location (placement in the annulus with no impedance on device function),
  * Intended performance of the prosthetic valve (aortic valve area > 1.2 cm2 for 26, 29 and 31mm valves, ≥ 0.9 cm2 for 23mm valve (by echocardiography using the continuity equation) and mean aortic valve gradient < 20 mmHg or peak velocity < 3 m/sec, without moderate or severe prosthetic valve aortic regurgitation)
  * Only one valve implanted in the proper anatomical location
Time Frame: Number of days from admission to discharge
Population: Participant Population= Consisted of all subjects with a TAVR index procedure who were evaluable for device success.
Measure: Number; unit: percentage of participants
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 468 | 141 | 378 | 0
percentage of participants | 84.6 | 88.7 | 86.8 |

19. Secondary Outcome: Procedural Success
Description: Medtronic CoreValve® System subjects only.
  Defined as device success and absence of in-hospital MACCE.
Time Frame: Number of days from admission to discharge
Population: Participant Population= Consisted of all subjects with a TAVR index procedure who were evaluable for procedural success.
Measure: Number; unit: percentage of participants
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 476 | 142 | 384 | 0
percentage of participants | 77.5 | 77.5 | 81.3 |

20. Secondary Outcome: Prosthetic Valve Dysfunction (PVD)
Description: PVD was defined according to VARC I using the Core Lab Echocardiography assessments including aortic regurgitation (AR) and aortic stenosis (AS) evaluations. Total AR reported as moderate or severe was considered PVD. AS was defined as significant stenosis and considered PVD if one of the following was met:
  * Peak velocity >4 m/s
  * Mean gradient >35 mmHg
  * EOA < 0.8 cm2
  * TVIV1 / TVIV2 < 0.25
Time Frame: 30 day, 6 month, 1 year, 2 year
Population: Participant Population= Consisted of all subjects with a valve implanted.
Measure: Number; unit: percentage of participants
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Number analyzed (Participants) | 486 | 148 | 390 | 354
percentage of participants
  30 day Aortic Stenosis | 2.3 | 6.1 | 3.1 | 4.8
  30 day Aortic Regurgitation | 23.5 | 16.9 | 13.6 | 1.7
  6 month Aortic Stenosis | 3.1 | 6.1 | 3.8 | 6.5
  6 month Aortic Regurgitation | 26.1 | 18.2 | 17.2 | 2.3
  1 year Aortic Stenosis | 3.5 | 6.1 | 4.9 | 8.2
  1 year Aortic Regurgitation | 27.0 | 19.6 | 17.9 | 2.8
  2 year Aortic Stenosis | 3.9 | 6.8 | 5.4 | 9.3
  2 year Aortic Regurgitation | 27.8 | 19.6 | 19.7 | 2.8

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from study enrollment to study closure, up to 5 years. Adverse event data are currently available and reported for up to 1 year
Description: All new or worsening AEs were collected through12 months.
Arm/Group | Extreme Risk: TAVI Iliofemoral | Extreme Risk: TAVI Non-Iliofemoral | High Risk: TAVI | High Risk: SAVR
Serious Adverse Events (participants affected / at risk) | 452/489 | 142/150 | 346/390 | 324/357
Other Adverse Events (participants affected / at risk) | 440/489 | 139/150 | 355/390 | 320/357
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extreme Risk: TAVI Iliofemoral (N=489) | Extreme Risk: TAVI Non-Iliofemoral (N=150) | High Risk: TAVI (N=390) | High Risk: SAVR (N=357)
Anaemia Deficiencies (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Anaemias Due To Chronic Disorders (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anaemias Haemolytic Immune (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemias Nec (Blood and lymphatic system disorders) | 140 (170) | 70 (75) | 106 (132) | 151 (173)
Coagulopathies (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 1 (1) | 4 (4)
Eosinophilic Disorders (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematological Disorders (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytoses Nec (Blood and lymphatic system disorders) | 5 (5) | 1 (1) | 3 (3) | 4 (4)
Marrow Depression And Hypoplastic Anaemias (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Thrombocytopenias (Blood and lymphatic system disorders) | 11 (11) | 4 (4) | 8 (8) | 22 (22)
Aortic Valvular Disorders (Cardiac disorders) | 44 (45) | 12 (12) | 42 (42) | 10 (12)
Cardiac Conduction Disorders (Cardiac disorders) | 106 (109) | 24 (27) | 79 (85) | 18 (19)
Cardiac Disorders Nec (Cardiac disorders) | 9 (9) | 3 (3) | 7 (9) | 7 (7)
Cardiac Signs And Symptoms Nec (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
Cardiac Valve Disorders Nec (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiomyopathies (Cardiac disorders) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Coronary Artery Disorders Nec (Cardiac disorders) | 6 (6) | 4 (4) | 9 (9) | 4 (4)
Heart Failures Nec (Cardiac disorders) | 117 (186) | 29 (43) | 69 (95) | 62 (85)
Ischaemic Coronary Artery Disorders (Cardiac disorders) | 28 (30) | 8 (8) | 15 (17) | 12 (15)
Mitral Valvular Disorders (Cardiac disorders) | 9 (9) | 5 (5) | 3 (3) | 5 (5)
Myocardial Disorders Nec (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Noninfectious Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pericardial Disorders Nec (Cardiac disorders) | 5 (7) | 4 (4) | 5 (5) | 10 (10)
Rate And Rhythm Disorders Nec (Cardiac disorders) | 28 (29) | 6 (6) | 16 (18) | 19 (19)
Right Ventricular Failures (Cardiac disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (1)
Supraventricular Arrhythmias (Cardiac disorders) | 65 (79) | 17 (22) | 43 (46) | 69 (80)
Tricuspid Valvular Disorders (Cardiac disorders) | 2 (2) | 3 (3) | 0 (0) | 2 (2)
Ventricular Arrhythmias And Cardiac Arrest (Cardiac disorders) | 48 (59) | 26 (30) | 27 (29) | 27 (27)
Cardiac Septal Defects Congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coagulation Disorders Congenital (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Male Reproductive Tract Disorders Congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vascular Anomalies Congenital Nec (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hearing Losses (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear Disorders Nec (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inner Ear Signs And Symptoms (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Thyroid Neoplasms (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blindness (Excl Colour Blindness) (Eye disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Cataract Conditions (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Corneal Infections, Oedemas And Inflammations (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lacrimal Disorders (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal Bleeding And Vascular Disorders (Excl Retinopathy) (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Retinal Structural Change, Deposit And Degeneration (Eye disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Retinal, Choroid And Vitreous Infections And Inflammations (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual Disorders Nec (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Abdominal Wall Conditions Nec (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Acute And Chronic Pancreatitis (Gastrointestinal disorders) | 4 (4) | 0 (0) | 2 (2) | 1 (1)
Anal And Rectal Ulcers And Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign Neoplasms Gastrointestinal (Excl Oral Cavity) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Excl Infective) (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 4 (4)
Diaphragmatic Hernias (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Excl Infective) (Gastrointestinal disorders) | 4 (4) | 3 (3) | 3 (3) | 2 (2)
Diverticula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Duodenal And Small Intestinal Stenosis And Obstruction (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2) | 3 (3)
Duodenal Ulcers And Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dyspeptic Signs And Symptoms (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Faecal Abnormalities Nec (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Flatulence, Bloating And Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastric And Oesophageal Haemorrhages (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric Ulcers And Perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Gastritis (Excl Infective) (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (2)
Gastrointestinal And Abdominal Pains (Excl Oral And Throat) (Gastrointestinal disorders) | 13 (15) | 4 (4) | 3 (3) | 2 (2)
Gastrointestinal Atonic And Hypomotility Disorders Nec (Gastrointestinal disorders) | 3 (3) | 1 (1) | 3 (4) | 1 (1)
Gastrointestinal Fistulae (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Necrosis And Gangrene (Excl Gangrenous Hernia) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Disorders Nec (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Signs And Symptoms Nec (Gastrointestinal disorders) | 15 (15) | 7 (7) | 7 (7) | 12 (13)
Gastrointestinal Spastic And Hypermotility Disorders (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Stenosis And Obstruction Nec (Gastrointestinal disorders) | 5 (5) | 1 (1) | 3 (3) | 3 (3)
Gastrointestinal Ulcers And Perforation, Site Unspecified (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Vascular Occlusion And Infarction (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Haemorrhoids And Gastrointestinal Varices (Excl Oesophageal) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Inguinal Hernias (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intestinal Haemorrhages (Gastrointestinal disorders) | 4 (4) | 1 (1) | 5 (5) | 4 (4)
Intestinal Ulcers And Perforation Nec (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Nausea And Vomiting Symptoms (Gastrointestinal disorders) | 2 (2) | 1 (2) | 3 (5) | 5 (5)
Non-Site Specific Gastrointestinal Haemorrhages (Gastrointestinal disorders) | 35 (40) | 18 (20) | 27 (29) | 16 (17)
Oesophageal Stenosis And Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oesophageal Ulcers And Perforation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Oesophagitis (Excl Infective) (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral Soft Tissue Pain And Paraesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic Neoplasms (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritoneal And Retroperitoneal Disorders (Gastrointestinal disorders) | 1 (2) | 2 (2) | 0 (0) | 2 (2)
Peritoneal And Retroperitoneal Haemorrhages (Gastrointestinal disorders) | 5 (5) | 1 (1) | 2 (2) | 1 (1)
Umbilical Hernias (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Administration Site Reactions Nec (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthenic Conditions (General disorders) | 11 (12) | 3 (3) | 9 (10) | 9 (9)
Body Temperature Altered (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cardiac Complications Associated With Device (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Complications Associated With Device Nec (General disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Death And Sudden Death (General disorders) | 10 (10) | 5 (5) | 6 (6) | 3 (3)
Device Issues Nec (General disorders) | 40 (40) | 7 (7) | 28 (30) | 2 (2)
Device Malfunction Events Nec (General disorders) | 1 (1) | 1 (1) | 5 (5) | 5 (5)
Febrile Disorders (General disorders) | 3 (3) | 2 (2) | 7 (7) | 6 (6)
Feelings And Sensations Nec (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Gait Disturbances (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
General Signs And Symptoms Nec (General disorders) | 7 (7) | 2 (2) | 4 (4) | 5 (5)
Healing Abnormal Nec (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hernias Nec (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Implant And Catheter Site Reactions (General disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Inflammations (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection Site Reactions (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mass Conditions Nec (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema Nec (General disorders) | 6 (7) | 1 (1) | 6 (7) | 6 (6)
Pain And Discomfort Nec (General disorders) | 26 (33) | 9 (11) | 23 (29) | 19 (22)
Product Physical Issues (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Therapeutic And Nontherapeutic Responses (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Withdrawal And Rebound Effects (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile Duct Infections And Inflammations (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis And Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 1 (1) | 4 (4) | 1 (1)
Hepatic And Hepatobiliary Disorders Nec (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic Failure And Associated Disorders (Hepatobiliary disorders) | 3 (3) | 0 (0) | 1 (1) | 3 (3)
Hepatic Fibrosis And Cirrhosis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular Damage And Hepatitis Nec (Hepatobiliary disorders) | 5 (5) | 0 (0) | 0 (0) | 2 (2)
Anaphylactic Responses (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal And Gastrointestinal Infections (Infections and infestations) | 6 (8) | 1 (1) | 4 (4) | 4 (4)
Atypical Mycobacterial Infections (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial Infections Nec (Infections and infestations) | 22 (25) | 6 (6) | 15 (20) | 12 (12)
Bone And Joint Infections (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Candida Infections (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Infections (Infections and infestations) | 6 (7) | 1 (1) | 1 (1) | 3 (3)
Central Nervous System And Spinal Infections (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Clostridia Infections (Gastrointestinal disorders) | 9 (9) | 2 (2) | 6 (7) | 6 (6)
Ear Infections (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterobacter Infections (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Enterococcal Infections (Infections and infestations) | 4 (5) | 0 (0) | 0 (0) | 2 (2)
Escherichia Infections (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fungal Infections Nec (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Haemophilus Infections (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes Viral Infections (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Infections Nec (Infections and infestations) | 8 (8) | 2 (2) | 6 (6) | 8 (8)
Infectious Transmissions (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza Viral Infections (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Klebsiella Infections (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lower Respiratory Tract And Lung Infections (Infections and infestations) | 74 (95) | 25 (26) | 44 (48) | 36 (43)
Pseudomonal Infections (Infections and infestations) | 1 (2) | 1 (1) | 1 (1) | 2 (2)
Sepsis, Bacteraemia, Viraemia And Fungaemia Nec (Infections and infestations) | 32 (35) | 17 (18) | 32 (38) | 29 (36)
Staphylococcal Infections (Infections and infestations) | 3 (3) | 4 (4) | 3 (3) | 3 (4)
Streptococcal Infections (Infections and infestations) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Upper Respiratory Tract Infections (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Urinary Tract Infections (Infections and infestations) | 28 (32) | 9 (11) | 21 (21) | 20 (22)
Vascular Infections (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral Infections Nec (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anaesthetic Complications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac And Vascular Procedural Complications (Injury, poisoning and procedural complications) | 16 (17) | 3 (4) | 7 (7) | 3 (3)
Cardiovascular Injuries (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Cerebral Injuries Nec (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 5 (5) | 2 (2)
Chest And Lung Injuries Nec (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fractures And Dislocations Nec (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 1 (1) | 3 (3)
Gastrointestinal And Hepatobiliary Procedural Complications (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Limb Injuries Nec (Incl Traumatic Amputation) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lower Limb Fractures And Dislocations (Injury, poisoning and procedural complications) | 18 (19) | 1 (1) | 9 (10) | 10 (12)
Non-Site Specific Injuries Nec (Injury, poisoning and procedural complications) | 13 (13) | 4 (4) | 14 (16) | 6 (6)
Non-Site Specific Procedural Complications (Injury, poisoning and procedural complications) | 25 (27) | 6 (6) | 25 (26) | 28 (29)
Pelvic Fractures And Dislocations (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
Poisoning And Toxicity (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Radiation Injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Reproductive System And Breast Injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory Tract And Thoracic Cavity Procedural Complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Site Specific Injuries Nec (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Skin Injuries Nec (Injury, poisoning and procedural complications) | 10 (11) | 1 (1) | 5 (5) | 5 (5)
Skin Procedural Complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skull Fractures, Facial Bone Fractures And Dislocations (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Spinal Fractures And Dislocations (Injury, poisoning and procedural complications) | 6 (7) | 1 (1) | 5 (8) | 2 (2)
Thoracic Cage Fractures And Dislocations (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Transfusion Related Complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Upper Limb Fractures And Dislocations (Injury, poisoning and procedural complications) | 10 (11) | 0 (0) | 2 (2) | 5 (6)
Bacteria Identification And Serology (Excl Mycobacteria) (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Counts Nec (Investigations) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Blood Gas And Acid Base Analyses (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Carbohydrate Tolerance Analyses (Incl Diabetes) (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cardiac Function Diagnostic Procedures (Investigations) | 2 (2) | 3 (3) | 0 (0) | 6 (6)
Coagulation And Bleeding Analyses (Investigations) | 5 (5) | 2 (2) | 6 (6) | 6 (7)
Ecg Investigations (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Liver Function Analyses (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Metabolism Tests Nec (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Microbiology And Serology Tests Nec (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Mineral And Electrolyte Analyses (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Physical Examination Procedures (Investigations) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Platelet Analyses (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Protein Analyses Nec (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Red Blood Cell Analyses (Investigations) | 13 (13) | 4 (4) | 10 (10) | 11 (11)
Renal Function Analyses (Investigations) | 4 (4) | 1 (1) | 2 (2) | 1 (1)
Respiratory Tract And Thoracic Imaging Procedures (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skeletal And Cardiac Muscle Analyses (Investigations) | 4 (4) | 2 (2) | 1 (1) | 5 (5)
Tissue Enzyme Analyses Nec (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinalysis Nec (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Function Analyses Nec (Investigations) | 3 (3) | 2 (2) | 0 (0) | 3 (3)
Vascular Tests Nec (Incl Blood Pressure) (Investigations) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
White Blood Cell Analyses (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appetite Disorders (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Calcium Metabolism Disorders (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (2)
Diabetes Mellitus (Incl Subtypes) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic Complications Dermal (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic Complications Nec (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Disorders Of Purine Metabolism (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Electrolyte Imbalance Nec (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 1 (1) | 1 (1)
General Nutritional Disorders Nec (Metabolism and nutrition disorders) | 18 (20) | 7 (7) | 4 (4) | 15 (16)
Hyperglycaemic Conditions Nec (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 3 (3) | 6 (6)
Hypoglycaemic Conditions Nec (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 3 (3) | 4 (4)
Magnesium Metabolism Disorders (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Metabolic Acidoses (Excl Diabetic Acidoses) (Metabolism and nutrition disorders) | 3 (3) | 3 (4) | 1 (1) | 4 (4)
Metabolic Alkaloses (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mixed Acid-Base Disorders (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Potassium Imbalance (Metabolism and nutrition disorders) | 14 (15) | 2 (2) | 8 (8) | 5 (6)
Protein Metabolism Disorders Nec (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sodium Imbalance (Metabolism and nutrition disorders) | 8 (10) | 2 (3) | 5 (5) | 5 (5)
Total Fluid Volume Decreased (Metabolism and nutrition disorders) | 15 (15) | 8 (8) | 8 (9) | 14 (15)
Total Fluid Volume Increased (Metabolism and nutrition disorders) | 12 (13) | 1 (1) | 7 (7) | 11 (12)
Arthropathies Nec (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Bone Disorders Nec (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone Related Signs And Symptoms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint Related Signs And Symptoms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 1 (1)
Metabolic Bone Disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle Weakness Conditions (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Musculoskeletal And Connective Tissue Pain And Discomfort (Musculoskeletal and connective tissue disorders) | 8 (9) | 1 (1) | 13 (15) | 7 (7)
Musculoskeletal And Connective Tissue Signs And Symptoms Nec (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myopathies (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Osteoarthropathies (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 3 (4) | 1 (1)
Spine And Neck Deformities (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
B-Cell Lymphomas Nec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Bladder Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Breast And Nipple Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Colonic Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gastric Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal Neoplasms Malignancy Unspecified Nec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Leukaemias Acute Myeloid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Multiple Myelomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myelodysplastic Syndromes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neoplasms Malignant Site Unspecified Nec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 2 (2) | 2 (2)
Neuromas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic Neoplasms Malignant (Excl Islet Cell And Carcinoid) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pharyngeal And Laryngeal Neoplasms Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatic Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Renal Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory Tract And Pleural Neoplasms Malignant Cell Type Unspecified Nec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Skin Neoplasms Malignant And Unspecified (Excl Melanoma) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Thyroid Neoplasms Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute Polyneuropathies (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Central Nervous System Haemorrhages And Cerebrovascular Accidents (Nervous system disorders) | 28 (28) | 14 (14) | 26 (30) | 32 (35)
Central Nervous System Vascular Disorders Nec (Nervous system disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Cerebellar Coordination And Balance Disturbances (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Coma States (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cortical Dysfunction Nec (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dementia (Excl Alzheimer's Type) (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Disturbances In Consciousness Nec (Nervous system disorders) | 9 (9) | 4 (5) | 14 (15) | 7 (8)
Dyskinesias And Movement Disorders Nec (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathies Nec (Nervous system disorders) | 14 (14) | 0 (0) | 4 (4) | 5 (5)
Encephalopathies Toxic And Metabolic (Nervous system disorders) | 8 (11) | 0 (0) | 3 (3) | 2 (2)
Headaches Nec (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hydrocephalic Conditions (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Increased Intracranial Pressure Disorders (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar Spinal Cord And Nerve Root Disorders (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Memory Loss (Excl Dementia) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Migraine Headaches (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mononeuropathies (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Nervous System Disorders Nec (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurological Signs And Symptoms Nec (Nervous system disorders) | 7 (8) | 8 (8) | 2 (2) | 11 (11)
Neuromuscular Junction Dysfunction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paralysis And Paresis (Excl Cranial Nerve) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Peripheral Neuropathies Nec (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizures And Seizure Disorders Nec (Nervous system disorders) | 3 (3) | 3 (4) | 1 (1) | 10 (10)
Sensory Abnormalities Nec (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Speech And Language Abnormalities (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Transient Cerebrovascular Events (Nervous system disorders) | 7 (8) | 1 (1) | 6 (6) | 2 (2)
Tremor (Excl Congenital) (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vagus Nerve Disorders (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety Symptoms (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Behaviour And Socialisation Disturbances (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion And Disorientation (Psychiatric disorders) | 6 (6) | 1 (1) | 8 (9) | 4 (4)
Deliria (Psychiatric disorders) | 3 (3) | 1 (1) | 4 (4) | 1 (1)
Depressive Disorders (Psychiatric disorders) | 3 (3) | 0 (0) | 2 (2) | 2 (2)
Mental Disorders Nec (Psychiatric disorders) | 13 (13) | 3 (4) | 4 (4) | 14 (14)
Perception Disturbances (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Suicidal And Self-Injurious Behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder And Urethral Symptoms (Renal and urinary disorders) | 7 (7) | 8 (9) | 8 (9) | 9 (11)
Bladder Disorders Nec (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Genital And Urinary Tract Disorders Nec (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephritis Nec (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephropathies And Tubular Disorders Nec (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Renal Disorders Nec (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal Failure And Impairment (Renal and urinary disorders) | 90 (108) | 31 (43) | 38 (42) | 58 (66)
Renal Failure Complications (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal Lithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal Obstructive Disorders (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal Vascular And Ischaemic Conditions (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Ureteric Disorders Nec (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Abnormalities (Renal and urinary disorders) | 10 (13) | 1 (1) | 8 (8) | 6 (11)
Breast Disorders Nec (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic Prolapse Conditions (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatic Neoplasms And Hypertrophy (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Reproductive Tract Disorders Nec (Excl Neoplasms) (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal Disorders Nec (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal Disorders Nec (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breathing Abnormalities (Respiratory, thoracic and mediastinal disorders) | 26 (27) | 21 (29) | 30 (33) | 26 (31)
Bronchial Conditions Nec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Bronchospasm And Obstruction (Respiratory, thoracic and mediastinal disorders) | 25 (28) | 16 (21) | 13 (15) | 8 (9)
Conditions Associated With Abnormal Gas Exchange (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1) | 6 (6) | 6 (6)
Coughing And Associated Symptoms (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 5 (6) | 0 (0)
Diaphragmatic Disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Laryngeal And Adjacent Sites Disorders Nec (Excl Infections And Neoplasms) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laryngeal Spasm, Oedema And Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower Respiratory Tract Inflammatory And Immunologic Conditions (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 6 (6) | 7 (7) | 8 (8)
Lower Respiratory Tract Signs And Symptoms (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mediastinal Disorders (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Nasal Disorders Nec (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1) | 5 (5) | 1 (1)
Parenchymal Lung Disorders Nec (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 3 (3) | 4 (4)
Pharyngeal Disorders (Excl Infections And Neoplasms) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax And Pleural Effusions Nec (Respiratory, thoracic and mediastinal disorders) | 54 (74) | 26 (36) | 29 (39) | 67 (86)
Pulmonary Hypertensions (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 5 (5) | 0 (0)
Pulmonary Oedemas (Respiratory, thoracic and mediastinal disorders) | 23 (24) | 3 (3) | 9 (9) | 10 (10)
Pulmonary Thrombotic And Embolic Conditions (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (1) | 1 (1) | 0 (0)
Respiratory Failures (Excl Neonatal) (Respiratory, thoracic and mediastinal disorders) | 54 (62) | 28 (29) | 36 (40) | 54 (68)
Respiratory Tract Disorders Nec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Tracheal Disorders (Excl Infections And Neoplasms) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Signs And Symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bullous Conditions (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dermal And Epidermal Conditions Nec (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dermatitis And Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dermatitis Ascribed To Specific Agent (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Purpura And Related Conditions (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rashes, Eruptions And Exanthems Nec (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin And Subcutaneous Tissue Ulcerations (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Skin Haemorrhages (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Injuries And Mechanical Dermatoses (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 6 (6) | 4 (4)
Skin Preneoplastic Conditions Nec (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Housing Circumstances (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Device Therapeutic Procedures (Surgical and medical procedures) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Corneal And Scleral Therapeutic Procedures (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fracture Treatments (Excl Skull And Spine) (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hernia Repairs (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Joint Therapeutic Procedures (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lens Therapeutic Procedures (Surgical and medical procedures) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Limb Therapeutic Procedures (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle Therapeutic Procedures (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prophylactic Procedures Nec (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Therapeutic Procedures (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Therapeutic Procedures Nec (Surgical and medical procedures) | 9 (9) | 0 (0) | 3 (3) | 2 (2)
Tracheal Therapeutic Procedures (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ureteric Therapeutic Procedures (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accelerated And Malignant Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Aneurysms And Dissections Non-Site Specific (Vascular disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
Aortic Aneurysms And Dissections (Vascular disorders) | 4 (4) | 3 (3) | 1 (1) | 5 (5)
Aortic Necrosis And Vascular Insufficiency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arterial And Aortic Injuries (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood Pressure Disorders Nec (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Circulatory Collapse And Shock (Vascular disorders) | 6 (7) | 2 (2) | 2 (2) | 4 (4)
Haemorrhages Nec (Vascular disorders) | 20 (24) | 13 (13) | 19 (19) | 10 (11)
Lymphangiopathies (Vascular disorders) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Lymphoedemas (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-Site Specific Embolism And Thrombosis (Vascular disorders) | 6 (7) | 1 (1) | 1 (1) | 2 (2)
Non-Site Specific Necrosis And Vascular Insufficiency Nec (Vascular disorders) | 3 (3) | 2 (2) | 3 (3) | 3 (3)
Non-Site Specific Vascular Disorders Nec (Vascular disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Peripheral Aneurysms And Dissections (Vascular disorders) | 5 (5) | 0 (0) | 9 (9) | 1 (1)
Peripheral Embolism And Thrombosis (Vascular disorders) | 21 (22) | 5 (5) | 7 (7) | 5 (6)
Peripheral Vascular Disorders Nec (Vascular disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Peripheral Vasoconstriction, Necrosis And Vascular Insufficiency (Vascular disorders) | 16 (18) | 2 (2) | 12 (12) | 2 (3)
Site Specific Vascular Disorders Nec (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 6 (7)
Varicose Veins Non-Site Specific (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular Hypertensive Disorders Nec (Vascular disorders) | 11 (11) | 3 (3) | 14 (15) | 7 (7)
Vascular Hypotensive Disorders (Vascular disorders) | 52 (54) | 15 (15) | 21 (23) | 38 (40)
Vascular Malformations And Acquired Anomalies (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extreme Risk: TAVI Iliofemoral (N=489) | Extreme Risk: TAVI Non-Iliofemoral (N=150) | High Risk: TAVI (N=390) | High Risk: SAVR (N=357)
Anaemias Nec (Blood and lymphatic system disorders) | 90 (98) | 27 (28) | 76 (77) | 69 (78)
Leukocytoses Nec (Blood and lymphatic system disorders) | 38 (42) | 18 (19) | 25 (26) | 46 (49)
Thrombocytopenias (Blood and lymphatic system disorders) | 68 (73) | 32 (33) | 61 (64) | 90 (95)
Cardiac Conduction Disorders (Cardiac disorders) | 114 (137) | 32 (37) | 80 (100) | 54 (68)
Heart Failures Nec (Cardiac disorders) | 30 (32) | 9 (9) | 20 (22) | 21 (24)
Rate And Rhythm Disorders Nec (Cardiac disorders) | 29 (30) | 12 (13) | 21 (22) | 30 (31)
Supraventricular Arrhythmias (Cardiac disorders) | 60 (66) | 36 (42) | 59 (69) | 80 (91)
Ventricular Arrhythmias And Cardiac Arrest (Cardiac disorders) | 31 (33) | 8 (10) | 22 (22) | 9 (9)
Gastrointestinal Atonic And Hypomotility Disorders Nec (Gastrointestinal disorders) | 36 (37) | 12 (12) | 22 (22) | 24 (24)
Nausea And Vomiting Symptoms (Gastrointestinal disorders) | 26 (33) | 7 (7) | 23 (25) | 16 (21)
Febrile Disorders (General disorders) | 36 (39) | 7 (8) | 16 (16) | 16 (16)
Oedema Nec (General disorders) | 44 (48) | 16 (18) | 34 (35) | 26 (31)
Pain And Discomfort Nec (General disorders) | 30 (34) | 9 (10) | 26 (30) | 30 (33)
Lower Respiratory Tract And Lung Infections (Infections and infestations) | 26 (26) | 16 (16) | 18 (19) | 21 (23)
Urinary Tract Infections (Infections and infestations) | 75 (80) | 28 (34) | 51 (59) | 58 (67)
Non-Site Specific Injuries Nec (Injury, poisoning and procedural complications) | 25 (26) | 2 (2) | 21 (23) | 11 (15)
Non-Site Specific Procedural Complications (Injury, poisoning and procedural complications) | 21 (23) | 6 (6) | 20 (21) | 29 (29)
Skeletal And Cardiac Muscle Analyses (Investigations) | 16 (16) | 7 (7) | 15 (15) | 19 (19)
Hyperglycaemic Conditions Nec (Metabolism and nutrition disorders) | 22 (22) | 6 (6) | 19 (19) | 29 (30)
Magnesium Metabolism Disorders (Metabolism and nutrition disorders) | 17 (17) | 9 (10) | 6 (6) | 9 (9)
Potassium Imbalance (Metabolism and nutrition disorders) | 56 (63) | 16 (25) | 36 (38) | 33 (37)
Sodium Imbalance (Metabolism and nutrition disorders) | 25 (26) | 10 (13) | 22 (22) | 28 (29)
Total Fluid Volume Increased (Metabolism and nutrition disorders) | 20 (20) | 12 (13) | 21 (21) | 41 (43)
Musculoskeletal And Connective Tissue Pain And Discomfort (Musculoskeletal and connective tissue disorders) | 34 (42) | 16 (19) | 34 (39) | 22 (22)
Neurological Signs And Symptoms Nec (Nervous system disorders) | 18 (20) | 2 (2) | 21 (22) | 17 (21)
Anxiety Symptoms (Psychiatric disorders) | 25 (25) | 6 (6) | 14 (14) | 14 (14)
Confusion And Disorientation (Psychiatric disorders) | 32 (34) | 13 (14) | 24 (25) | 23 (25)
Renal Failure And Impairment (Renal and urinary disorders) | 67 (78) | 16 (20) | 40 (43) | 44 (51)
Breathing Abnormalities (Respiratory, thoracic and mediastinal disorders) | 26 (26) | 8 (8) | 27 (29) | 14 (16)
Bronchospasm And Obstruction (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 10 (11) | 4 (5) | 10 (10)
Conditions Associated With Abnormal Gas Exchange (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 8 (11) | 11 (12) | 11 (11)
Parenchymal Lung Disorders Nec (Respiratory, thoracic and mediastinal disorders) | 35 (35) | 10 (10) | 23 (23) | 41 (41)
Pneumothorax And Pleural Effusions Nec (Reproductive system and breast disorders) | 76 (82) | 30 (32) | 52 (58) | 91 (105)
Pulmonary Oedemas (Respiratory, thoracic and mediastinal disorders) | 29 (29) | 5 (5) | 20 (20) | 26 (27)
Haemorrhages Nec (Vascular disorders) | 34 (35) | 4 (4) | 26 (26) | 9 (9)
Vascular Hypertensive Disorders Nec (Vascular disorders) | 45 (49) | 20 (20) | 46 (55) | 37 (40)
Vascular Hypotensive Disorders (Vascular disorders) | 68 (73) | 18 (21) | 40 (41) | 40 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less